CLINICAL TRIAL: NCT01133639
Title: Does Ketorolac Delay Bone Healing and Improve Post-operative Pain?: A Prospective Double-Blind Placebo-Controlled Randomized Clinical Trial
Brief Title: Ketorolac Effects on Post-operative Pain and Bone Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer with the institution, funding issues, poor accrual
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American College of Foot and Ankle Surgeons (Other)
Responsible Party: Principal Investigator, Emily Cook, Instructor in Surgery, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P000047
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Bunion
MeSH Terms: conditions — Bunion | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo plus standard of care
  Interventions: Drug: Placebo
- Ketorolac (Experimental): 30 mg IV dose intra-operatively followed by 10 mg orally every 8 hours for five days plus standard of care
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — 30 mg IV dose intra-operatively followed by 10 mg orally every 8 hours for five days plus standard of care
  Arms: Ketorolac
Drug: Placebo — Placebo plus standard of care
  Arms: Placebo

SUMMARY:
This will be a randomized double-blind placebo-controlled clinical trial that will accept all eligible consecutive patients undergoing elective Kalish bunionectomies. Patients will be randomized into either receiving ketorolac (30 mg IV dose intra-operatively followed by 10 mg orally every 8 hours for five days) plus standard of care or placebo plus standard of care. The purpose of this study is to evaluate the effects of ketorolac plus standard of care on post-operative pain control and radiographic osseous healing. Patients will be assessed for pain via a validated pain questionnaire and for delayed unions via a radiographic scoring system shown to have both high inter- and intra-observer reliability by a blinded board certified radiologist. Additional outcomes of bunionectomy procedures will also be evaluated including adverse events and time to regular shoe gear and activities.

ELIGIBILITY:
Inclusion Criteria:

* Hallux abductus with bunion deformity
* Adult patients as defined by >=18 years old and <= 65 years old
* Subject has adequate perfusion, verified by the surgeon, which is defined by palpable pedal pulses
* Subject has voluntarily signed and dated an informed consent form, approved by IRB, and provided HIPAA (or other applicable privacy regulation) authorization prior to any participation in the study
* Subject agrees not to take any new medications, dietary supplements, or alternative therapies during the study period (approximately 12 weeks)
* Subject is interested in participating in the study and willing to comply with the study protocol
* Patient has pain related to a bunion deformity but pain-free metatarsalphalangeal joint (MTPJ) range of motion that is not functionally adapted
* Adequate bone density to withstand a Kalish bunionectomy procedure
* No frontal plane hallux deformity
* Minimal abnormality of the PASA
* Normal to minimally malaligned sagittal plane position of the first metatarsal
* Failure of conservative treatment
* General Pre-operative Radiographic Angle Criteria† - 10-15 degree IMA in rectus feet* - 20-25 degree TAA in adducted feet* - 15-20 degree IMA in rectus feet if wide metatarsal head width - 25-30 degree TAA in adducted feet if wide metatarsal head width IMA=intermetatarsal angle; TAA=total adductus angle *If the pre-operative IMA is <15 degree, only the IMA will be used pre-operatively. For IMA >=15, the total adductus angle will be used †These are general guidelines and the width of the metatarsal as well as the presence of positional, structural, or combined first ray deformity may also influence procedure selection.

Exclusion Criteria:

* a history of an allergic-type reaction in response to exposure to aspirin, phenylacetic acid derivatives, or other NSAIDs
* hypersensitivity to ketorolac tromethamine, or to any product component
* any known bleeding risk or bleeding disorder, suspected or confirmed
* history of or active cerebrovascular bleeding, suspected or confirmed
* concomitant aspirin or NSAID use where the patient may not be advised to discontinue the medication during the study
* concomitant pentoxifylline use
* concomitant probenecid use
* coronary artery bypass graft (CABG) surgery within one year of the procedure
* any history of gastrointestinal bleeding/perforation, gastrointestinal ulcer, severe peptic ulcer disease, or severe inflammatory bowel disease
* hemorrhagic diathesis, suspected or confirmed
* incomplete intraoperative hemostasis
* pre-operative serum creatinine > 1.5 ml/dL or blood urea nitrogen level > 22 mg/dL
* any history of renal impairment or risk of renal failure due to volume depletion

  * Patients with a known allergy, contraindication and/or intolerance for oxycodone 5mg - acetaminophen 325 mg will be excluded from the study.
  * Patients with a known allergy, contraindication, and/or intolerance for the local anesthetic (bupivicaine) or any of the standardized intra-operative opioids and anti-emetics administered by the anesthesiologist
  * Patients with a history of fibromyalgia or opioid abuse
  * History of chronic regional pain syndrome or diagnosis of any chronic pain syndrome, patients requiring routine methadone or other opioids
  * Neuropathy or radiculopathy
  * Subject has alcohol or substance abuse, dementia, brain metastases, or other cognitive disorders that may interfere with pain assessment and the post-operative course outlined by the surgeon
* American Society of Anesthesiologists (ASA) Physical Status class four or higher
* women who are pregnant, planning on becoming pregnant, or breast feeding
* presence of active local or systemic infection
* subject has a myocardial infarction in the last twelve months

  • Patients who are not candidates for a Kalish bunionectomy due to the preoperative deformity as well as other study exclusions are:
* Absent pedal pulses or ABI < 0.9 and > 1.2
* Concomitant midfoot and rearfoot procedures
* Moderate to high abnormal PASA angles
* Significant sagittal plane first metatarsal deformity
* Moderate to severe osteoporosis as evaluated by preoperative radiographs and/or bone mineral density tests
* Revision cases
* History of previous infections, radiation treatment, or current infection related to the surgical site
* History of previous trauma of the first metatarsal or first ray
* Subject has known immunosuppression (HIV, recent chemotherapy, organ transplant)
* Patients taking systemic steroid (patients taking less than 5 mg of prednisone, inhaled steroids for asthma or chronic obstructive pulmonary disease, topical or optical steroids will not be excluded)
* Subject has active malignancy, excluding cutaneous malignancies except melanoma Pregnancy Elective bunion surgery will not be performed if the patient is pregnant or planning on becoming pregnant during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Cook, DPM, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 subjects were enrolled & completed the study. Pharmacy held the randomization table. PI left institution & was never unblinded (because there were never any AEs). Therefore, do not know which subjects were in the placebo vs ketorolac arms. Study was terminated due to lack of administrative support 2/2012 & all data has been destroyed.
Period: Overall Study
Arm/Group | Placebo | Ketorolac
Started (See comments in Recruitment Details section above. Maximum length is too short to explain here.) | 0 (18 total subjects were enrolled, study was terminated prematurely and data was not analyzed) | 0 (18 total subjects were enrolled, study was terminated prematurely and data was not analyzed)
Completed (See comments in Recruitment Details section above. Maximum length is too short to explain here.) | 0 (18 total subjects were enrolled, study was terminated prematurely and data was not analyzed) | 0 (18 total subjects were enrolled,study was terminated prematurely and data was not analyzed)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 18 subjects were enrolled & completed the study. Pharmacy held the randomization table. PI left institution & was never unblinded (b/c there were never any AEs). Therefore, do not know which subjects were in the placebo vs ketorolac arms. Study was terminated due to lack of administrative support 2/2012 & all data has been destroyed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ketorolac | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Pain
Description: 18 subjects were enrolled & completed the study. Pharmacy held the randomization table. PI left institution & was never unblinded (because there were never any AEs). Therefore, do not know which subjects were in the placebo vs ketorolac arms. Study was terminated due to lack of administrative support 2/2012 & all data has been destroyed.
Time Frame: Post-Operative Day 2
Population: 18 subjects were enrolled & completed the study. Pharmacy held the randomization table. PI left institution & was never unblinded (because there were never any AEs). Therefore, do not know which subjects were in the placebo vs ketorolac arms. Study was terminated due to lack of administrative support 2/2012 & all data has been destroyed.
Arm/Group | Placebo | Ketorolac
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Osseous Healing
Description: Radiographic assessment by a blinded board certified radiologist
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Placebo | Ketorolac
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Post-operative Activity Recovery
Description: Functional Recovery Index
Time Frame: up to 3 months
Population: as for outcome 1
Arm/Group | Placebo | Ketorolac
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adverse Events
Description: Comparison of adverse events between the two study arms
Time Frame: 1 week
Population: as for outcome 1
Arm/Group | Placebo | Ketorolac
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quantity of Narcotic Medication
Description: Comparison of quantity of narcotic medication utilized within the two study arms
Time Frame: 1 week
Population: as for outcome 1
Arm/Group | Placebo | Ketorolac
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 subjects were enrolled & all subjects completed the study. Adverse events were monitored & assessed through study completion for each subject. Pharmacy held the randomization table. Per study protocol, any adverse event would have required unblinding of the PI & reporting to the IRB. PI left institution & was never unblinded (b/c there were never any AEs). Therefore, do not know which subjects were in the placebo vs ketorolac arms. But no adverse events occurred with any of the subjects.
Description: Pharmacy maintained the randomization table. The PI was blinded as she was also one of the surgeons in the study. The PI left the institution & was never unblinded or given the randomization table because there were never any adverse events & the data was never analyzed. PI terminated the study due to lack of administrative support. Study terminated 2/2012 & data has been destroyed and was never analyzed. Do not know which subjects were in placebo vs ketorolac arm.
Groups:
- Placebo or Ketorolac: Placebo: Placebo plus standard of care
  or
  Ketorolac 30 mg IV dose intra-operatively followed by 10 mg orally every 8 hours for five days plus standard of care
  Ketorolac: 30 mg IV dose intra-operatively followed by 10 mg orally every 8 hours for five days plus standard of care
Arm/Group | Placebo or Ketorolac
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-04-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT01133639/Prot_SAP_001.pdf